CLINICAL TRIAL: NCT03827876
Title: An Open-Label Study Evaluating Enstilar® (Calcipotriene and Betamethasone Dipropionate) Foam, 0.005%/0.064% QD in Psoriasis Patients Being Treated With Etanercept or Adalimumab
Brief Title: Enstilar in Combination With Enbrel or Humira for Plaque Psoriasis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC04
Record Dates: First submitted 2019-01-29; First posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Intervention Model Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label Enstilar (Experimental): once daily for 4 weeks followed by QOD for 12 weeks for patients receiving Enbrel or Humira
  Interventions: Drug: Enstilar 0.005%-0.064% Topical Foam

INTERVENTIONS:
Drug: Enstilar 0.005%-0.064% Topical Foam — Enstilar 0.005%-0.064% Topical Foam applied once daily for 4 weeks followed by QOD for 12 weeks for patients receiving Enbrel or Humira

SUMMARY:
4 weeks of adjunctive therapy of Enstilar® QD followed by 12 weeks QOD to patients with 2-10% BSA who are receiving etanercept or adalimumab for at least 24 weeks

DETAILED DESCRIPTION:
30 subjects treated with etanercept or adalimumab for at least 24 weeks with a body surface area 2-10% and physician global assessment greater than or equal to 2 will receive Enstilar® once daily for 4 weeks followed by QOD for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult ≥ 18 years of age;
* Diagnosis of chronic plaque-type
* Patient with 2-10% BSA
* Physician Global Assessment of 2 or greater
* Patient has been treated with etanercept or adalimumab for a minimum of 24 weeks

Exclusion Criteria:

* ˂2 or >10% BSA
* PGA <2
* Patient not receiving etanercept or adalimumab, or receiving etanercept or adalimumab <24weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-09-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
PGA x BSA improvement | 16 weeks
  body surface area multiplied by physician global assessment

SECONDARY OUTCOMES:
BSA improvement | 16 weeks
  body surface area improvement
Dermatology Life Quality Index improvement | 16 weeks
  patient reported outcome improvements of DLQI (Dermatology Life Quality Index). Calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired. The DLQI can also be expressed as a percentage of the maximum possible score of 30.
Itch Numerical Rating Scale | 16 weeks
  Patient reported itch scale from 0 (no itch) to 10 (worst imaginable itch).

CONTACTS AND LOCATIONS:
Locations (1):
- Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No